CLINICAL TRIAL: NCT02193152
Title: A Pilot Study of Pazopanib in Molecularly Selected Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Pazopanib in Molecularly Selected Patients With Advanced NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated by sponsor
Sponsor: Washington University School of Medicine (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201408009
Record Dates: First submitted 2014-07-11; First posted 2014-07-17 (Estimated); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Carcinoma, Non-Small Cell Lung; Non-Small Cell Lung Cancer; Nonsmall Cell Lung Cancer
Keywords: Advanced Non-Small Cell Lung Cancer; NSCLC; Pazopanib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment: Pazopanib (Experimental): Pazopanib 800 mg daily should be taken orally without food at least one hour before or two hours after a meal.
  One cycle of pazopanib is 28 days.
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib
  Other Names: GW786034; Votrient®

SUMMARY:
The purpose of this study is to evaluate how participants with advanced non-small cell lung cancer (NSCLC) that have certain abnormalities in the pazopanib target genes respond to pazopanib treatment.

DETAILED DESCRIPTION:
There has been a limited benefit from anti-angiogenesis drugs in patients with NSCLC. Bevacizumab provides a modest survival improvement when added to chemotherapy and VEGFR tyrosine kinase inhibitors have been associated with minimal efficacy as single agents and increased toxicity when combined with chemotherapy. We postulate that the response rates and survival may be improved with a better selection of patients based on abnormalities of the targets for the drugs. According to the preliminary data from the cancer genome atlas (TCGA), the targets of pazopanib are altered in 28% of patients with adenocarcinoma and 24% of patients with squamous cell lung cancer. Since, despite the molecular selection prior to treatment, only a small percentage of patients will benefit from the treatment, we plan to further investigate those patients with whole exome sequencing in both the pre-treatment samples to identify the predictors for response and at the time of progression, with repeated biopsy, in an attempt to identify the predictors for secondary resistance. By identifying more reliable predictors for response to pazopanib, our study may help to establish its role in the treatment of NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of advanced (metastatic or unresectable) non-small cell lung cancer (NSCLC) with mutations, rearrangement and fusion involving RET oncogene, or abnormalities in the pazopanib target genes defined as VEGFR1-3, PDGFRA, PDGFRB, or TP53 with abnormalities including deletion, insertion, early stop codon, and/or nonsynonymous mutations with functional consequences. CLIA certified lab testing for pazopanib target genes using cell free DNA from peripheral blood and/or assays performed on tumor tissues are acceptable.
* Evaluable disease by imaging or physical exam OR measurable disease defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* Failed at least one standard chemotherapeutic treatment for NSCLC.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Hemoglobin ≥ 9.0 g/dL
  * PT or INR ≤ 1.2 x IULN
  * aPTT ≤ 1.2 x IULN
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN
  * Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 30 mL/min/1.73 m2 for patients with creatinine levels above 1.5 mg/dL
  * UPC < 1 or, if UPC ≥ 1, 24-hour urine protein < 1 g; use of urine dipstick for renal function assessment is not acceptable.
* Patients receiving anticoagulation therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation.
* Ability to swallow and retain oral tablets.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Treatment with any of the following anti-cancer therapies:

  * Radiation therapy, surgery, or tumor embolization within 14 days prior to the first dose of pazopanib OR
  * Chemotherapy, immunotherapy, investigational therapy or hormonal therapy within 14 days prior to the first dose of pazopanib
* Prior treatment with any VEGFR tyrosine kinase inhibitor.
* Administration of any non-oncologic investigational drug within 30 days or 5 half-lives (whichever is longer) prior to the first dose of pazopanib.
* Use of a strong CYP3A4 inhibitor less than 14 days prior to initiation of study treatment
* A history of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Symptomatic brain metastases. Patients with known brain metastases are allowed if they are asymptomatic.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to pazopanib or other agents used in the study.
* Any ongoing toxicity from prior anti-cancer therapy that is > grade 1 and/or that is progressing in severity (except alopecia). Any IO related adverse events must be ≤ grade 1 to be eligible.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled seizure disorder, chronic underlying liver disease unrelated to cancer, or psychiatric illness/social situations that would limit compliance with study requirements.
* Corrected QT interval (QTc) > 480 msecs.
* History of any one or more of the following cardiovascular conditions within the past 6 months: cardiac angioplasty or stenting, myocardial infarction, unstable angina pectoris, coronary artery bypass graft surgery, symptomatic peripheral vascular disease, class III or IV congestive heart failure as defined by the New York Heart Association (see Appendix B).
* Poorly controlled hypertension (defined as systolic blood pressure of ≥ 140 mmHg or diastolic blood pressure of ≥ 90 mmHg). Note: initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. Following antihypertensive medication initiation or adjustment, blood pressure must be reassessed three times at approximately 2-minute intervals. At least 24 hours must have elapsed between antihypertensive medication initiation or adjustment and blood pressure measurement. These three values should be averaged to obtain the mean diastolic and systolic blood pressures, which must be < 140/90 mmHg in order for a patient to be eligible for the study.
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding, including (but not limited to) active peptic ulcer disease, known intraluminal metastatic lesions with risk of bleeding, inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease) or other GI conditions with increased risk of perforation, history of abdominal fistula or intra-abdominal abscess within 28 days prior to beginning study treatment.
* Clinically significant gastrointestinal abnormalities that may affect absorption of pazopanib, including (but not limited to) malabsorption syndrome or major resection of the stomach or small bowel.
* History of cerebrovascular accident including transient ischemic attack, pulmonary embolism (including asymptomatic or previously treated PE), or untreated deep venous thrombosis within the past 6 months. Patients with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible.
* Major surgery or trauma within 28 days prior to first dose of pazopanib and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major surgery).
* Evidence of active bleeding or bleeding diathesis.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage. Note: lesions infiltrating major pulmonary vessels (contiguous tumor and vessels) are excluded; however, the presence of a tumor that is touching but not infiltrating (abutting) the vessels is acceptable (CT with contrast is strongly recommended to evaluate such lesions). Large protruding endobronchial lesions in the mail or lobar bronchi are excluded; however, endobronchial lesions in the segmented bronchi are allowed. Lesions extensively infiltrating the main or lobar bronchi are excluded; however, minor infiltrations in the wall of thee bronchi are allowed.
* Recent hemoptysis (≥ ½ teaspoon of red blood within 8 weeks before first dose of pazopanib).
* Pregnant and/or breastfeeding. Patient must have a negative serum pregnancy test within 14 days of study entry.
* Known HIV-positivity. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2019-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Morgensztern, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment: Pazopanib
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment: Pazopanib
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 66.5 [50 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: * Participants should be re-evaluated for response 8 weeks after initiation of pazopanib and then every 8 weeks thereafter. In addition to a baseline scan, confirmatory scans should also be obtained not less than 4 weeks following initial documentation of objective response.
  * Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) [Eur J Ca 45:228-247, 2009].
  * Response rate is the percentage of participants with a complete or partial response
  * Complete response=Disappearance of all target and non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
  * Partial response=At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters
Time Frame: Until the end of treatment (median length of treatment=85.5 days (full range 25-334 days)
Population: 4 participants were not evaluable for this outcome measure because they were removed from treatment prior to the re-evaluation response at 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: Pazopanib
Number analyzed (Participants) | 12
Participants | 2

2. Primary Outcome: Progression-free Survival (PFS)
Description: * Progression-free survival is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. There is no limit on following for progression-free survival besides death of the participant.
  * Progressive disease=At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: Until progressive disease or death (median follow-up 174 days, full range 41 days-545 days)
Measure: Median (Full Range); unit: weeks
Arm/Group | Treatment: Pazopanib
Number analyzed (Participants) | 16
weeks | 13.25 [3.5 to 47.8]

3. Secondary Outcome: Outcomes Associated With Specific Mutations
Description: * Participants are followed until death.
  * All participants will undergo next generation sequencing prior to enrollment into the study.
  * Initial predictors are the mutations in VEGFR or PDGFR, but sequencing will be used to evaluate for other predictors as well.
Time Frame: Until time of death (an expected average of 8 months)
Population: The data was not collected for this outcome measure.
Arm/Group | Treatment: Pazopanib
Number analyzed (Participants) | 0

4. Secondary Outcome: Mutational Predictors for Extreme Responders
Description: -Whole exome and transcriptome sequencing will be performed in 10 participants, including 4 to 6 responders and 4 to 6 non-responders in order to identify the predictors for benefit.
Time Frame: Until end of treatment (an expected average of 8 months)
Population: The data was not collected for this outcome measure.
Arm/Group | Treatment: Pazopanib
Number analyzed (Participants) | 0

5. Secondary Outcome: Mechanisms of Secondary Resistance.
Description: -Participants will also undergo next generation sequencing at the time of progression in an attempt to identify the mechanisms for secondary resistance.
Time Frame: Until the time of progressive disease (an expected average of 8 months)
Population: The data was not collected for this outcome measure.
Arm/Group | Treatment: Pazopanib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from study start through 30 days after completion of treatment (median treatment length 85.5 days (full range=25 days-334 days)).
Arm/Group | Treatment: Pazopanib
All-Cause Mortality (participants affected / at risk) | 14/16
Serious Adverse Events (participants affected / at risk) | 8/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment: Pazopanib (N=16)
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Lung infection (Infections and infestations) | 3
Upper respiratory infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Death (Investigations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Syncope (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment: Pazopanib (N=16)
Anemia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Visual changes (Eye disorders) | 1
Hypothryoidism (Endocrine disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 7
Gingival pain (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 5
Chills (General disorders) | 6
Dry mouth (General disorders) | 1
Edema limbs (General disorders) | 7
Edema face (General disorders) | 2
Fatigue (General disorders) | 14
Leg pain (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Foot pain (General disorders) | 1
Left side pain (General disorders) | 1
Fever (General disorders) | 2
Flu like symptoms (General disorders) | 2
Hip pain (General disorders) | 1
Shoulder pain (General disorders) | 1
Papulopustular rash (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Infection (Infections and infestations) | 3
Platelet count decreased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 2
Creatinine increased (Investigations) | 1
Weight loss (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 10
Hypercalcemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Left shoulder pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 10
Headache (Nervous system disorders) | 9
Peripheral sensory neuropathy (Nervous system disorders) | 12
Memory impairment (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 12
Confusion (Psychiatric disorders) | 3
Polyuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 6
Bruising (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Nail changes (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 4
Palmar-plantar erythrodysethesia (Skin and subcutaneous tissue disorders) | 2
Hot flashes (Vascular disorders) | 6
Hypertension (Vascular disorders) | 9
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT02193152/Prot_SAP_000.pdf